CLINICAL TRIAL: NCT04777617
Title: Assessment of Donor Derived Cell-free DNA in Combined Kidney-pancreas Recipients
Brief Title: Allosure in Simultaneous Pancreas Kidney Transplant
Status: Terminated | Type: Observational
Why Stopped: slow enrollment
Sponsor: Washington University School of Medicine (Other)
Collaborators: CareDx (Industry); University of Texas (Other)
Responsible Party: Sponsor
Other Study IDs: 202011048
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Kidney Pancreas Transplant
Keywords: Kidney pancreas transplant; Deceased donor cell free DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WU/Barnes cohort: SPK patients in this group will be recruited from WU/Barnes Transplant center. A total of 25 from this cohort will be recruited and asked to provide a blood sample to test for donor derived cell free DNA 3 times over the course of the first year of transplant. In addition, if any biopsies or rejections occur, additional samples will be requested at the time of biopsy and for an additional two follow-ups at least one month apart.
  Interventions: Other: DD-cfDNA
- UT Southwestern cohort: SPK patients in this group will be recruited from WU/Barnes Transplant center. A total of 25 from this cohort will be recruited and asked to provide a blood sample to test for donor derived cell free DNA 3 times over the course of the first year of transplant. In addition, if any biopsies or rejections occur, additional samples will be requested at the time of biopsy and for an additional two follow-ups at least one month apart.
  Interventions: Other: DD-cfDNA

INTERVENTIONS:
Other: DD-cfDNA — We are obtaining samples for donor derived cell free DNA in an observational manner. There is no intervention in this study

SUMMARY:
This study will observe donor derived cell free DNA percentages (via the Allosure test) in combined kidney-pancreas transplant recipients to establish both stable and dysfunctional Allosure assay levels

DETAILED DESCRIPTION:
Simultaneous kidney-pancreas transplantation is the optimal treatment for select patients with type 1 diabetes and kidney failure. Limited biomarkers are utilized to monitor the health of the allografts. For kidney transplantation serum creatinine remains the most commonly monitored biomarker; for the pancreas allograft blood glucose and serum amylase and lipase are measured. However, these biomarkers are imprecise and non-specific for rejection.

In kidney transplantation cell free donor derived DNA at of value of >1% has emerged as an effective immune monitoring tool as a marker for renal allograft rejection and injury. Thus far, a discriminatory donor derived cell free DNA value for a stable and rejecting allografts has not been established for recipients of combined kidney-pancreas transplants.

Study aim will be to help establish a normal range of donor derived cell free DNA in stable kidney-pancreas graft function in combined kidney pancreas transplant recipients while determining changes in cell free DNA in kidney-pancreas recipients with biopsy proven allograft rejection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Kidney-pancreas transplant recipients
* Patient must have stable creatine, lipase, amylase for at least a two month span after transplant OR patient must receive a biopsy within one year post transplant

Exclusion Criteria:

* Presence of non-renal or pancreas transplanted organ
* Patient is not enrolled within 1 year after transplant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This population will be SPK patients with stable Cr, lipase and amylase for at least 2 months post transplant and enrolled within the first year after transplant
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
DD-cfDNA level | 1 year
  determine level of donor derived cell free DNA from SPK patients

CONTACTS AND LOCATIONS:
Overall Officials: Rowena Delos Santos, MD, Principal Investigator — Washington University in Saint Louis School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bloom RD, Bromberg JS, Poggio ED, Bunnapradist S, Langone AJ, Sood P, Matas AJ, Mehta S, Mannon RB, Sharfuddin A, Fischbach B, Narayanan M, Jordan SC, Cohen D, Weir MR, Hiller D, Prasad P, Woodward RN, Grskovic M, Sninsky JJ, Yee JP, Brennan DC; Circulating Donor-Derived Cell-Free DNA in Blood for Diagnosing Active Rejection in Kidney Transplant Recipients (DART) Study Investigators. Cell-Free DNA and Active Rejection in Kidney Allografts. J Am Soc Nephrol. 2017 Jul;28(7):2221-2232. doi: 10.1681/ASN.2016091034. Epub 2017 Mar 9. PMID 28280140
- [Background] Grskovic M, Hiller DJ, Eubank LA, Sninsky JJ, Christopherson C, Collins JP, Thompson K, Song M, Wang YS, Ross D, Nelles MJ, Yee JP, Wilber JC, Crespo-Leiro MG, Scott SL, Woodward RN. Validation of a Clinical-Grade Assay to Measure Donor-Derived Cell-Free DNA in Solid Organ Transplant Recipients. J Mol Diagn. 2016 Nov;18(6):890-902. doi: 10.1016/j.jmoldx.2016.07.003. Epub 2016 Oct 7. PMID 27727019